CLINICAL TRIAL: NCT04007445
Title: Exercise Training in a Community-based Setting for People with Spinal Cord Injuries
Brief Title: Exercise for People with Spinal Cord Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: The Craig H. Neilsen Foundation (Other)
Responsible Party: Principal Investigator, Kerri Morgan, Assistant Professor of Occupational Therapy and Neurology, Washington University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 201701143
Record Dates: First submitted 2019-07-01; First posted 2019-07-05 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2020-05

CONDITIONS: Spinal Cord Injuries
Keywords: spinal cord injury; exercise; occupational therapy
MeSH Terms: conditions — Spinal Cord Injuries; Motor Activity | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: The proposed project utilizes a mixed methods approach. An experimental strategy using a randomized control trial (single-blinded) will be used to assess the efficacy of an established transitional, community-based exercise intervention on people with SCI. Qualitative methods will be used to gather information related to optimizing implementation of a community-based exercise intervention. This project will be conducted in conjunction with Paraquad, a local independent living center. Forty participants will be randomized into an Exercise Group (EG) or Control Group (CG) by the statistician who will not be involved in either conducting outcome assessments or implementation of the intervention. This design will assist in reducing variability and maximizing the effect size for powering subsequent larger randomized control trials.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Formally Directed Group (Exercise Group) (Active Comparator): A group performing a 12 - week guided exercise program at an accessible Community Health and Wellness Center
  Interventions: Behavioral: Formally Directed Group (Exercise Group)
- Self-Directed Group (Control Group) (Placebo Comparator): A group receiving educational information about physical activity and exercise at home and then self-directing a 12 - week exercise program on their own.
  Interventions: Other: Self-Directed Group (Control Group)

INTERVENTIONS:
Behavioral: Formally Directed Group (Exercise Group) — This group will receive a 12-week exercise intervention that will educate and support the person's ability to exercise. Working with a trainer, the participant will attend a 12-week (3 x week) exercise program that has been personalized to their goals. Each session will include warm-up, stretching, cardiovascular exercises, strength exercises, and cool-down. Each session will be 1-2 hours in duration. The participants may wear accelerometers and heart rate monitors to help determine the level of intensity of the exercises, as they should be performing at least 150 minutes of moderate to vigorous exercise each week. By the end of the 12-week program, the goal is for participants to guide their own exercise regimens.
  Arms: Formally Directed Group (Exercise Group)
Other: Self-Directed Group (Control Group) — This group will receive a 1-hour education session during which they will learn about the National Council on Health, Physical Activity and Disability (NCHPAD) website, an information and resource center on health promotion for people with disabilities. During the session participants will be given an overview of the website and asked to find three resources they find of interest. Their strength and fitness will also be assessed by completing a 1-rep max test. The participants will then be asked to maintain their regular physical activity for the next 12 weeks and complete a weekly physical activity log to track their exercise participation. A staff member will phone each person every week for the 12-week period and have the participant report his or her physical activity during the week.
  Arms: Self-Directed Group (Control Group)

SUMMARY:
The purpose of the study is to examine the impact of a transitional exercise intervention implemented in the community for people with SCI on psychological well-being, social factors, and physiological health.

DETAILED DESCRIPTION:
People with spinal cord injuries (SCI) are at a greater risk for major health conditions and poorer health outcomes than the population without disabilities. For people with SCI, physical activity is critical for both physiological and psychological well-being. Currently a gap exists; prior research indicates that exercise programs conducted in a controlled clinical setting have positive effects on the physical and psychosocial fitness of people with SCI, but rarely are these programs available in accessible community-based exercise facilities. With this study, the investigators aim to evaluate the improvements of the exercise group - EG (formally-directed) in both psychological and physiological well-being as compared to the control group - CG (self-directed). The investigators also aim to identify the perspectives of the participants on the recruitment and enrollment process, the assessment methods, and the intervention protocol. The long-term goal of this research is to improve outcomes of people with SCI once they leave rehabilitation by identifying strategies to promote health and support exercise in the community. This study will implement rigorous research procedures to examine a transitional exercise intervention in the community for people with SCI. This study will serve as the initial step toward that goal by pilot testing an exercise intervention to help with the transition from supported exercise programs experienced during rehabilitation to the community. The investigators will recruit 40 adults with SCI to participate in this study; the EG will participate in a transitional 12-week exercise intervention at Paraquad Health and Wellness Center (PQHWC). The CG will participate in a one-hour education session, learning about the National Council on Health, Physical Activity and Disability (NCHPAD), and then they will maintain their typical physical activity on their own for a 12-week period. This project will measure the potential psychosocial and physiological health benefits of participating in a transitional community-based exercise intervention. The investigators will then use the findings to define how exercise in the community can support health outcomes and improve therapeutic interventions to promote health of people with SCI.

ELIGIBILITY:
Inclusion Criteria:

Participants will be non-exercising adults with SCI who have participated in less than 60 minutes of moderate-intensity exercise per week in the last month. Participants must meet the following inclusion criteria: diagnosis of an SCI; are 18 years or older; have written physician approval to participate in the study; have the ability to use upper, lower, or both sets of extremities to exercise; and have the ability to understand English.

Exclusion Criteria:

Participants will be excluded if they are medically unstable, have a cognitive impairment that does not allow them to provide consent, are currently or have previously been participants in the PQHWC or community-based exercise program, or have been enrolled in a structured exercise program over the past six months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2020-04-29 (Actual); Study Completion 2020-04-29 (Actual)

PRIMARY OUTCOMES:
PROMIS - Change in Fatigue (Short Form 8a) | Baseline, post intervention and 3 month follow-up
  The Fatigue item banks assess a range of self-reported symptoms, from mild subjective feelings of tiredness to an overwhelming, debilitating, and sustained sense of exhaustion that likely impacts one's ability to execute daily activities and function normally in family or social roles. Fatigue is divided into the experience of fatigue and the impact of fatigue. The fatigue short forms are not disease specific and assess fatigue over the past seven days. PROMIS instruments are scored using item-level calibrations. Each question is answered using a 5-point Likert scale from "not at all (1)" to "very much (5)". Calculate a summed score and then use the applicable PROMIS score conversion table to translate the total raw score into a T-score.
  The seven domains are scored individually, and the single pain intensity item is reported as its raw score.
PROMIS - Change in Emotional Distress - Depression (Short Form 8a) | Baseline, post intervention and 3 month follow-up
  The Depression item banks assess self-reported negative mood (sadness, guilt), views of self(self-criticism, worthlessness), and social cognition (loneliness, interpersonal alienation), as well as changed positive affect and engagement (loss of interest, meaning, and purpose). The depression short forms are not disease specific and assess depression over the past seven days. PROMIS instruments are scored using item-level calibrations. Each question is answered using a 5-point Likert scale from "never (1)" to "always (5)". Calculate a summed score and then use the applicable PROMIS score conversion table to translate the total raw score into a T-score.
  The seven domains are scored individually, and the single pain intensity item is reported as its raw score.
PROMIS - Change in Pain Intensity (Short Form 3a) | Baseline, post intervention and 3 month follow-up
  The Pain Intensity instruments assess how much a person hurts. The pain intensity short forms are not disease specific and assess pain intensity over the past seven days. PROMIS instruments are scored using item-level calibrations. Each question is answered using a 5-point Likert scale from "Had no pain (1)" to "very severe (5)". Calculate a summed score and then use the applicable PROMIS score conversion table to translate the total raw score into a T-score.
  The seven domains are scored individually, and the single pain intensity item is reported as its raw score.
PROMIS - Change in Pain Interference (Short Form 8a) | Baseline, post intervention and 3 month follow-up
  The Pain Interference item banks assess self-reported consequences of pain on relevant aspects of one's life. This includes the extent to which pain hinders engagement with social, cognitive, emotional, physical, and recreational activities. It also incorporates items probing sleep and enjoyment in life. The pain interference short forms are not disease specific and assess pain interference over the past seven days. PROMIS instruments are scored using item-level calibrations. Each question is answered using a 5-point Likert scale from "not at all (1)" to "very much (5)". Calculate a summed score and then use the applicable PROMIS score conversion table to translate the total raw score into a T-score.
  The seven domains are scored individually, and the single pain intensity item is reported as its raw score.
PROMIS - Change in Sleep Disturbance (Short Form 8a) | Baseline, post intervention and 3 month follow-up
  The Sleep disturbance instruments assess self-reported perceptions of sleep quality, sleep depth, and restoration associated with sleep. This includes perceived difficulties and concerns with getting to sleep or staying asleep, as well as perceptions of the adequacy of and satisfaction with sleep. The sleep disturbance short forms are not disease specific and assess sleep disturbances over the past seven days. PROMIS instruments are scored using item-level calibrations. Each question is answered using a 5-point Likert scale from "very poor (1)" to "very good (5)". Calculate a summed score and then use the applicable PROMIS score conversion table to translate the total raw score into a T-score.
  The seven domains are scored individually, and the single pain intensity item is reported as its raw score.
PROMIS - Change in Emotional Support | Baseline, post intervention and 3 month follow-up
  The Emotional support item banks assess perceived feelings of being cared for and valued as a person; having confident relationships. PROMIS instruments are scored using item-level calibrations. Each question is answered using a 5-point Likert scale from "never (1)" to "always (5)". Calculate a summed score and then use the applicable PROMIS score conversion table to translate the total raw score into a T-score.
  The seven domains are scored individually, and the single pain intensity item is reported as its raw score.

SECONDARY OUTCOMES:
The Exercise Self-Efficacy Scale (ESES) | Baseline, post intervention, 3 month follow-up
  The ESES is a 10-item, SCI-specific scale developed to measure perceived exercise self-efficacy for various types of physical activities. The scale requires individuals to self-report their confidence in performing physical activities and exercise. One dichotomous item asks whether the individual has exercised at home and/or in a gym in the past 12 months. Individuals respond to the 10 items using a four-point Likert scale (1: not at all true, 4: always true); the total score is then derived by summing the scores for the individual items; scores range from 10 to 40. Higher scores indicate greater perceived self-efficacy. The dichotomous item is used to estimate the participant's average exercise activity.
RM 4-FM: Motivation for Physical Activity and Exercise/Working Out - Questionnaire | Baseline, post intervention, 3-month follow-up
  The RM 4-FM assesses a person's motivation for exercise or working out to determine the impact of intrinsic and extrinsic factors.

CONTACTS AND LOCATIONS:
Overall Officials: Kerri A Morgan, PhD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gray DB, Hollingsworth HH, Stark SL, Morgan KA. Participation survey/mobility: psychometric properties of a measure of participation for people with mobility impairments and limitations. Arch Phys Med Rehabil. 2006 Feb;87(2):189-97. doi: 10.1016/j.apmr.2005.09.014. PMID 16442971
- [Background] Miller LC, Gottlieb M, Morgan KA, Gray DB. Interviews with employed people with mobility impairments and limitations: environmental supports impacting work acquisition and satisfaction. Work. 2014;48(3):361-72. doi: 10.3233/WOR-131784. PMID 24284677
- [Background] Kroll T, Kehn M, Ho PS, Groah S. The SCI Exercise Self-Efficacy Scale (ESES): development and psychometric properties. Int J Behav Nutr Phys Act. 2007 Aug 30;4:34. doi: 10.1186/1479-5868-4-34. PMID 17760999
- [Background] American College of Sports Medicine. (2010). ACSM's Guidelines for Exercise Testing and Prescription. 8th ed. Philadelphia: Lippincott Williams & Wilkins.
- [Background] Kroll T, Barbour R, Harris J. Using focus groups in disability research. Qual Health Res. 2007 May;17(5):690-8. doi: 10.1177/1049732307301488. PMID 17478650
- [Background] Krueger RA, Casey MA. (2009). Focus Groups: A Practical Guide For Applied Research 4th ed. Thousand Oaks, CA: Sage.
- [Background] White GW, Suchowierska M, Campbell M. Developing and systematically implementing participatory action research. Arch Phys Med Rehabil. 2004 Apr;85(4 Suppl 2):S3-12. doi: 10.1016/j.apmr.2003.08.109. PMID 15083417
- [Background] Askari S, Kirby RL, Parker K, Thompson K, O'Neill J. Wheelchair propulsion test: development and measurement properties of a new test for manual wheelchair users. Arch Phys Med Rehabil. 2013 Sep;94(9):1690-8. doi: 10.1016/j.apmr.2013.03.002. Epub 2013 Mar 14. PMID 23499781
- [Background] Ginis KA, Arbour-Nicitopoulos KP, Latimer AE, Buchholz AC, Bray SR, Craven BC, Hayes KC, Hicks AL, McColl MA, Potter PJ, Smith K, Wolfe DL. Leisure time physical activity in a population-based sample of people with spinal cord injury part II: activity types, intensities, and durations. Arch Phys Med Rehabil. 2010 May;91(5):729-33. doi: 10.1016/j.apmr.2009.12.028. PMID 20434610
- [Background] Jelleyman C, Yates T, O'Donovan G, Gray LJ, King JA, Khunti K, Davies MJ. The effects of high-intensity interval training on glucose regulation and insulin resistance: a meta-analysis. Obes Rev. 2015 Nov;16(11):942-61. doi: 10.1111/obr.12317. PMID 26481101
- [Background] Cowan RE, Callahan MK, Nash MS. The 6-min push test is reliable and predicts low fitness in spinal cord injury. Med Sci Sports Exerc. 2012 Oct;44(10):1993-2000. doi: 10.1249/MSS.0b013e31825cb3b6. PMID 22617394